CLINICAL TRIAL: NCT03912168
Title: Does Giving a Question Prompt List to Patients With Orthopaedic Conditions Improve Their Perceived Involvement in Care? A Randomized Controlled Trial
Brief Title: Question Prompt List for Orthopaedic Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robin Kamal, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 50238
Record Dates: First submitted 2019-04-08; First posted 2019-04-11 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Tendon Injuries; Fracture; Arthritis; Sprains; Strains; Tumor; Pain
MeSH Terms: conditions — Tendon Injuries; Fractures, Bone; Arthritis; Sprains and Strains; Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Question Prompt List (Experimental)
  Interventions: Other: Question Prompt List
- 3 questions list (Active Comparator)
  Interventions: Other: 3 questions list

INTERVENTIONS:
Other: Question Prompt List — Question prompt list for common orthopaedic conditions
  Arms: Question Prompt List
Other: 3 questions list — 3 questions from the AskShareKnow model
  Arms: 3 questions list

SUMMARY:
The purpose of this study is to investigate whether providing patients with a question prompt list (QPL) prior to their orthopaedic surgery clinic appointment improves their perceived involvement in care (PICs) score compared to being given 3 questions from the AskShareKnow model

ELIGIBILITY:
Inclusion Criteria:

* common orthopaedic condition new patient

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Perceived involvement in care scale | Immediately after the clinical encounter, same day as clinical encounter
  The Perceived involvement in care scale PICS measures a patient's perceived involvement in their visit. it is a 13 item validated scale, scored 0-13, with higher scores indicating greater perceived involvement

CONTACTS AND LOCATIONS:
Overall Officials: Robin N Kamal, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mariano DJ, Liu A, Eppler SL, Gardner MJ, Hu S, Safran M, Chou L, Amanatullah DF, Kamal RN. Does a Question Prompt List Improve Perceived Involvement in Care in Orthopaedic Surgery Compared with the AskShareKnow Questions? A Pragmatic Randomized Controlled Trial. Clin Orthop Relat Res. 2021 Feb 1;479(2):225-232. doi: 10.1097/CORR.0000000000001582. PMID 33239521